CLINICAL TRIAL: NCT01757860
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of CARD-024 (1α-Hydroxy-Vitamin-D5) in Healthy Subjects
Brief Title: Safety and Pharmacokinetics Study of CARD-024 in Healthy Subjects
Acronym: CARD-024
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardiavent Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARD-024-C001
Record Dates: First submitted 2012-12-17; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Drug Safety; Heart; Disease, Activity
MeSH Terms: conditions — Disease; Motor Activity | interventions — Drug Carriers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CARD-024 (Experimental): CARD-024 oral administered: 3, 9, 27 or 81 mcg.
  Interventions: Drug: CARD-024
- Drug Carrier (Placebo Comparator): Placebo: 20% ethanol:80% propylene glycol solution oral administered.
  Interventions: Other: Drug Carrier

INTERVENTIONS:
Drug: CARD-024 — Comparison of different dosages of drug
  Other Names: 1α-Hydroxy-Vitamin-D5; 1αVitD5
  Arms: CARD-024
Other: Drug Carrier — Drug Carrier, 20% ethanol:80% propylene glycol oral administered solution.
  Other Names: Placebo, Drug Carrier
  Arms: Drug Carrier

SUMMARY:
Study Phase: Phase 1

Primary Objective:

• To evaluate the safety and tolerability of single ascending oral doses of CARD-024 in healthy subjects

Secondary Objectives:

* To evaluate the pharmacokinetic (PK) profile of CARD-024 following ascending single oral doses of CARD-024
* To evaluate the effect of CARD-024 on cardiovascular indices including plasma renin activity (PRA) and blood pressure (BP), biological markers of activity, following ascending single oral doses of CARD-024

DETAILED DESCRIPTION:
Study Design: This is a single-center, double-blind, randomized, placebo-controlled study of single oral doses of CARD-024. Four planned cohorts of 8 subjects each will be dosed sequentially and randomized to receive a single dose of active drug (6 subjects) or placebo (2 subjects). Cohort 4 will have 10 subjects randomized to receive active drug (7 subjects) or placebo (3 subjects). Each cohort will be divided into at least 2 groups; the first group will have 2 subjects, 1 receiving active drug and 1 receiving placebo. Dosing of the remaining 6 subjects in each cohort will be completed in a manner agreed upon by the Sponsor and the Principal Investigator in keeping with the randomization schedule and blinded conditions.

The planned cohorts are:

Cohort CARD-024 Dose*

1. 3 μg
2. 9 μg
3. 27 μg
4. 81 μg

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between the ages of 18 and 55, inclusive, with body mass index (BMI) between 18-32 kg/m2.
2. Females must be surgically sterile or at least 2 years post-menopausal. Menopausal status will be verified by a follicular stimulating hormone (FSH) test. Those with bilateral tubal ligation must also use a barrier method of birth control. In addition, all females must have a negative pregnancy test at Screening.
3. No clinically significant findings on physical examination, including BP, pulse rate and 12-lead ECG. No clinically significant medical history.
4. No clinically significant safety laboratory results at Screening. Cardiavent, Inc. - CONFIDENTIAL
5. Nonsmoker or light smoker (≤5 cigarettes per day or similar use of other tobacco products) and are willing to refrain from smoking while in the clinic.
6. Willing and able to sign an informed consent document indicating understanding the purpose of and procedures required for the study and willingness to participate in the study.
7. Willing and able to stay in the clinic for the inpatient activities required by the protocol for all visits.

Exclusion Criteria:

1. Evidence of clinically relevant pathology that could interfere with the study results or put the subject's safety at risk.
2. Current or recurrent disease that may affect the action, absorption, or disposition of the study treatment, or clinical or laboratory assessments.
3. Current or relevant previous history of serious, severe, or unstable (acute or progressive) physical or psychiatric illness, any medical disorder requiring treatment or that may make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study treatment or procedures.
4. History of febrile illness within the 5 days prior to the first dose.
5. Positive Hepatitis B surface antigen (HbsAg), Hepatitis C antibody or Human Immunodeficiency Virus (HIV) test result at Screening visit.
6. Use of any prescription medication or over-the-counter (OTC) medication within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication or during the study. As an exception, acetaminophen may be used at doses up to 1 g/day.
7. Use of any herbal supplements (including herbal weight-loss or "metabolism booster" therapies) within 30 days prior to the first dose of trial medication.
8. Known or suspected intolerance or hypersensitivity to similar study drugs or excipients, closely related compounds or any of their stated ingredients.
9. Positive screen for alcohol or drugs of abuse during Screening visit or at study check-in for Day 1 dosing.
10. Participated in a clinical study involving an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to study drug administration.
11. Blood donation of 1 pint or more within 56 days of the start of the study.
12. Plasmapheresis or plasma donation within 30 days of the start of the study.
13. Single 12-lead ECG demonstrating QTc >450 msec at Screening, and or history or evidence of long QT syndrome. A single repeat ECG may be done at the Principal Investigator's discretion.
14. Any condition that in the opinion of the Principal Investigator would complicate or compromise the study or the well-being of the subject.
15. Unwilling or unable to comply with the clinic house rules.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety | 5 days
  Adverse events such as nausea, vomiting, headache, muscle ache, neuralgia and patient overall tolerance to drug.

SECONDARY OUTCOMES:
Drug Pharmacokinetics | 5 days
  Measure of drug absorption and elimination by measuring drug blood levels after oral administration. Assessment of drug C-max, T-lag, T-1/2, AUC, Vd/F and K-a.
Drug Pharmacodynamics | 5 days
  Measure of pharmacodynamics by 1] measuring plasma renin activity (PRA), 2] measuring plasma parathyroid hormone (PTH) levels, and 3] measuring drug effect on systolic and diastolic blood pressure by arm cuff occlusion.

OTHER OUTCOMES:
Induction of Hypercalcemia | 5 days
  Measure of serum calcium levels post treatment to assess drug calcemic activity.

CONTACTS AND LOCATIONS:
Overall Officials: James Vanderlugt, MD, Principal Investigator — Jasper Clinic, Michigan; Robert U Simpson, PhD, Study Chair — Cardiavent Inc.
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States